CLINICAL TRIAL: NCT03692312
Title: A Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Tideglusib Versus Placebo for the Treatment of Children and Adolescents With Congenital Myotonic Dystrophy (REACH CDM)
Brief Title: Efficacy and Safety of Tideglusib in Congenital Myotonic Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AMO Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMO-02-MD-2-003; 2016-004623-23 (EudraCT Number)
Expanded Access: NCT07119775 (Available)
Record Dates: First submitted 2018-03-16; First posted 2018-10-02 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Congenital Myotonic Dystrophy
Keywords: Tideglusib; AMO-02-MD-2-003; Congenital Myotonic Dystrophy; Myotonic Dystrophy; Dystrophia Myotonica; Myotonia Atrophica; Myotonia Dystrophica; Myotonic Dystrophy, Congenital; Steinert Disease; Steinert Myotonic Dystrophy; Steinert's Disease
MeSH Terms: conditions — Myotonic Dystrophy | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tideglusib (Experimental): Weight adjusted tideglusib, orally, once daily
  Interventions: Drug: Tideglusib; Drug: Placebo
- Placebo (Placebo Comparator): Matching placebo, orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tideglusib — Tideglusib for oral suspension, weight-adjusted at 400mg, 600mg or 1000 mg dose levels, once daily
  Arms: Tideglusib
Drug: Placebo — Matching placebo formulation

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled, Phase 2/3 study of patients (aged 6 to 16 years) diagnosed with Congenital Myotonic Dystrophy (Congenital DM1).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study of weight adjusted dose 1000 mg/day tideglusib versus placebo in the treatment of children and adolescents 6-16 years of age with Congenital DM1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children and adolescents aged ≥6 years and ≤16 years
2. Diagnosis of Congenital DM1 (also known as Steinert's disease)

   * Diagnosis must be genetically confirmed
   * One or more of the following clinically relevant (e.g. requiring medical intervention) signs or symptoms was evident within the first month after birth:

     * Hypotonia
     * Generalized weakness
     * Respiratory insufficiency
     * Feeding difficulties
     * Clubfoot or another musculoskeletal deformity
3. Subject must be able to walk and complete the 10-meter walk-run test (orthotics/splints allowed, forearm crutches are not allowed)
4. Written, voluntary informed consent must be obtained before any study related procedures are conducted.

   * Where a parent or LAR provides consent, there must also be assent from the subject
5. Subject's caregiver must be willing and able to support participation for duration of study
6. Subject must be willing and able to comply with the required food intake restrictions as outlined per protocol

Exclusion Criteria:

1. Not able to walk; (full time wheel chair use)
2. Body mass index (BMI) less than 13.5 kg/m² or greater than 40 kg/m²
3. New or change in medications/therapies within 4 weeks prior to Screening
4. Use of strong CYP3A4 inhibitors (e.g clarithromycin, telithromycin, ketoconazole, itraconazole, posaconazole, nefazodone, idinavir and ritonavir) within 4 weeks prior to Baseline
5. Concurrent use of drugs metabolized by CYP3A4 with a narrow therapeutic window (e.g. warfarin and digitoxin)
6. Current enrollment in a clinical trial of an investigational drug or enrollment in a clinical trial of an investigational drug in the last 6 months
7. Existing or historical medical conditions or complications (e.g. neurological, cardiovascular, renal, hepatic, endocrine, gastrointestinal or respiratory disease) which would cause the investigator to conclude that the subject will not be able to perform the study procedures or assessments or would confound interpretation of data obtained during assessment
8. Hypersensitivity to tideglusib and its excipients including allergy to strawberry

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Horrigan, MD, Study Director — AMO Pharma
Locations (14):
- United States (9):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Palo Alto, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Rochester Medical Center, Rochester, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University - Department of Neurology. Muscular Dystrophy Translational Research Program., Richmond, Virginia
- The Bright Alliance, Randwick, New South Wales, Australia
- Canada (2):
  - Children's Hospital London Health Sciences Centre (LHSC), London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- New Zealand Clinical Research (NZCR), Auckland, New Zealand
- Newcastle University, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children and adolescents (≥6 - ≤16 years) with a diagnosis of genetically confirmed congenital type 1 myotonic dystrophy. Subjects were to have a Clinical Global Impression-Severity score of ≥4 at Screening and V2, be ambulatory and able to complete the 10m walk/run test. Planned randomization of 56 subjects closed at 53 subjects due to fewer than expected discontinuations. A participant assigned to placebo was found to have some tideglusib levels and was included in analysis sets for tideglusib
Groups:
- Tideglusib: Weight adjusted tideglusib, orally, once daily
  Tideglusib for oral suspension, weight-adjusted at 400 mg for 2 weeks, then up-titrated to a weight-adjusted 600 mg for 2 weeks, after which 1000 mg was administered for the remainder of the treatment period, once daily
Period: Overall Study
Arm/Group | Tideglusib | Placebo
Started | 27 | 26
Completed | 25 | 25
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all randomized subjects who received at least one dose of study treatment. Subjects were presented by treatment actually received. A participant assigned to placebo was found to have some tideglusib levels (due to inadvertent exposure between siblings in opposing arms), and was therefore, included in the safety analysis and full analysis sets for tideglusib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tideglusib | Placebo | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.0 (3.32) | 11.0 (3.61) | 11.0 (3.43)
Age, Customized [Median (Full Range); unit: years]
  Median | 10 [6 to 16] | 11 [6 to 16] | 10 [6 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 19 | 16 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethic origin n (%): Hispanic or Latino | 3 | 5 | 8
  Ethic origin n (%): Not Hispanic or latino | 25 | 20 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race n (%): Black or African American | 0 | 1 | 1
  Race n (%): American Indian or Alaska Native | 1 | 0 | 1
  Race n (%): Asian | 0 | 2 | 2
  Race n (%): White | 27 | 18 | 45
  Race n (%): Other | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Completed Congenital DM1 Rating Scale (CDM1-RS)
Description: The Clinician-Completed Congenital DM1 Scale is an 11-item rating scale completed by the clinician that scores the symptom severity of domains that are clinically relevant in Congenital DM1.
  The severity of the clinician's concern in each domain is scored by using a 5-point Likert Scale. Scores range from 0 = Not present to 4 = Very severe.
Time Frame: Baseline and week 20
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 26
score on a scale | -1.65 (0.620) | -3.40 (0.618)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; Analysis is a mixed model for repeated measures (MMRM) analysis with treatment, visit, age group and treatment by visit interaction as fixed effects and baseline value as a covariate. An unstructured variance-covariance matrix has been used; Test type: Superiority; p = 0.0514, MMRM; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [-0.01 to 3.51], Standard Error of Mean 0.875

2. Secondary Outcome: Change in Clinical Global Impression- Improvement Scale (CGI-I) Scores
Description: The clinician administered CGI-I rates how much the subject's illness has improved or worsened relative to a baseline state.
  A 7-point Likert type scale is used with ratings of 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Baseline and week 20
Population: A subject (randomized to tideglusib) withdrew consent on Day 12 of randomized treatment and was excluded from the intent-to-treat analysis, full and per-protocol analysis sets as they did not have a post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 26 | 26
score on a scale | 3.11 (0.190) | 2.77 (0.189)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2124, MMRM; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.20 to 0.88], Standard Error of Mean 0.268

3. Secondary Outcome: Change in Top 3 Caregiver Concerns Visual Analogue Scale (VAS) Score
Description: The Top 3 concerns VAS allows caregivers to identify their main three causes of concern, related to the subject's myotonic dystrophy, rather than these being pre-specified within a scale and then rating how these concerns have changed at specific time-points during the study. Caregivers were asked to rate three causes for concern by drawing a vertical mark on a 10 cm long VAS with anchors of "not at all severe" at the left end (0 cm) and "very severe" at the right end (10 cm). A score for each concern was to be determined by measuring the number of centimeters on the 10 cm VAS line from the anchor point on the left side of the line. A total VAS score for each subject was calculated as the sum of the scores for the 3 concerns (minimum = 0 cm, maximum = 30 cm). A higher score represents a worse outcome.
Time Frame: Baseline and week 20
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | -1.74 (0.780) | -6.47 (0.780)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = 4.74, 95% CI 2-sided [2.51 to 6.96], Standard Error of Mean 1.104

4. Secondary Outcome: Caregiver Completed Congenital DM1 Rating Scale (CC-CDM1-RS)
Description: The Caregiver-Completed Congenital DM1 Scale is a caregiver assessment of the subject on symptoms that may occur in individuals with CDM1. There are a total of 11 clinically relevant symptoms that the caregiver is asked to rate the severity of.
  The symptoms are rated on a score from 0 to 4 based on overall severity where 0 = symptom not present or is no longer present during the relevant time frame, and 4 = very severe, symptom causes pronounced and consistent impairment and is highly disruptive with regard to daily life. A total CC-CDM1-RS score for each subject was calculated as the sum of the scores where 0 = min and 44 = max. A higher score represents a worse outcome.
Time Frame: Baseline and week 20
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | -0.18 (0.770) | -3.36 (0.782)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0059, MMRM; Mean Difference (Final Values) = 3.18, 95% CI 2-sided [0.96 to 5.39], Standard Error of Mean 1.099

5. Secondary Outcome: Clinical Global Impression - Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity Scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis.
  Subjects are assessed on severity of illness at the time of rating 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Baseline and week 20
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | -0.20 (0.076) | -0.12 (0.076)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4634, MMRM; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.30 to 0.14], Standard Error of Mean 0.108

6. Secondary Outcome: 10-meter Walk-run Test
Description: The 10-meter walk/run test is a performance measure used to assess walking speed in seconds over a short distance. It can be used as an assessment of functional mobility.
Time Frame: 20 weeks
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 25
Seconds | -0.54 (0.393) | -0.19 (0.391)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5385, MMRM; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.49 to 0.79], Standard Error of Mean 0.564

7. Secondary Outcome: Number of Adverse Events (AEs), Including Serious Adverse Events (SAEs), Between Screening to End of Study.
Description: Adverse events may be volunteered spontaneously by the subject, or discovered as a result of general, non-leading questioning by physician.
Time Frame: Between Screening to End of Study, up to 28 weeks
Population: A participant assigned to placebo was found to have some tideglusib levels (due to inadvertent exposure between siblings in opposing arms), and was therefore, included in the safety analysis and full analysis sets for tideglusib.
Measure: Count of Participants; unit: Participants
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 28 | 25
Participants
  Total number of TEAEs | 20 | 19
  Total number of serious TEAEs | 1 | 0
  Total number of serious TEAEs related to treatment | 0 | 0
  Total number of subjects with TEAEs leading to discontinuation from the study | 1 | 0
  Total number of subjects with treatment-related TEAEs leading to discontinuation from the study | 1 | 0
  Total number of subjects with TEAEs leading to death | 0 | 0
  Severity: Mild | 13 | 15
  Severity: Moderate | 7 | 4
  Severity: Severe | 0 | 0
  Unrelated to active treatment | 18 | 17
  Related to active treatment | 2 | 2

8. Secondary Outcome: Number of Abnormal Findings in Objective Assessments (e.g. Laboratory Values, ECGs, Vital Signs and Bone Mineral Density) Between Screening and End of Study.
Description: Abnormal laboratory findings (e.g. hematology, liver function, biochemistry, urinalysis) or other abnormal assessments (e.g. ECGs, vital signs) that are judged by the Investigator as clinically significant will be recorded as AEs or SAEs if they meet the definition of an AE. The Investigator will exercise his or her medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Time Frame: Between Screening to End of Study, up to 28 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 28 | 25
Participants
  Alanine aminotransferase increased | 1 | 0
  Haemoglobin decreased | 1 | 0
  Transaminases increased | 1 | 0
  Weight decreased | 0 | 2

9. Secondary Outcome: CDM1-RS Independent Central Rater Score (CDM1-RS)
Description: Change from baseline to end of treatment in the independent central rater CDM1-RS total score. CDM1 Rating Scale is an 11-item rating scale completed by the clinician to score the symptom severity that are clinically relevant in CDM1.
  The severity of the clinician's concern in each domain is scored by using a 5-point Likert Scale. Scores range from 0 = Not present to 4 = Very severe.
Time Frame: Baseline to week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Tideglusib: Weight adjusted tideglusib, orally, once daily
  Tideglusib for oral suspension, weight-adjusted at 400mg for 2 weeks, then up-titrated to a weight-adjusted 600mg for 2 weeks, after which 1000 mg was administered for the remainder of the treatment period, once daily
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 20 | 19
score on a scale | -2.26 (0.533) | -2.55 (0.547)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7110, MMRM; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.26 to 1.83], Standard Error of Mean 0.764

10. Secondary Outcome: CGI-I Independent Central Rater Score (CGI-I)
Description: The CGI-I requires the clinician to rate how much the subject's illness has changed (improved, worsened or stayed the same) relative to a baseline state on a seven point scale.
  A 7-point Likert type scale is used with ratings of 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Baseline and week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 25 | 23
score on a scale | 2.74 (0.227) | 2.65 (0.234)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7861, MMRM; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.57 to 0.75], Standard Error of Mean 0.326

11. Secondary Outcome: Independent Rater Clinical Global Impression - Severity Scale (CGI-S)
Description: CGI-S is a 7-point Likert type scale. An independent central rater rated the CGI-S scales for both the in-clinic and telehealth interviews.
  Subjects are assessed on severity of illness at the time of rating 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Baseline and week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 21 | 19
score on a scale | -0.15 (0.080) | -0.21 (0.093)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; Analysis is a mixed model for repeated measures (MMRM) analysis with treatment, visit, age group and treatment by visit interaction as fixed effects and baseline value as a covariate. A compound symmetry variance-covariance matrix has been used; Test type: Superiority; p = 0.6282, MMRM; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.19 to 0.31], Standard Error of Mean 0.123

12. Post Hoc Outcome: MDRI Analysis
Description: A multi-domain responder index (MDRI) analysis was performed by combining 5 endpoints to objectively assess movement, muscle integrity and strength, cognitive skills and adaptive behavior. For each of the 5 endpoints, subjects were scored +1 point if their change exceeded or was equal to the threshold in a beneficial direction, -1 point if their change exceeded or was equal to the threshold in a detrimental direction and 0 points otherwise. The sum of these 5 scores were added together to provide an MDRI score between -5 and 5, where a higher score indicates greater overall improvement.
Time Frame: Baseline and week 20
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 24 | 24
score on a scale | 0.8 (0.31) | -0.1 (0.25)
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; Test type: Superiority; p = 0.0428, t-test, 2 sided

13. Post Hoc Outcome: Creatine Phosphokinase
Description: Analysis of Ratio to Baseline in Creatine Phosphokinase
Time Frame: 20 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio to Baseline
Arm/Group | Tideglusib | Placebo
Number analyzed (Participants) | 24 | 24
Ratio to Baseline | 0.81 [0.68 to 0.97] | 1.05 [0.89 to 1.26]
Statistical Analysis 1: Comparison: Tideglusib vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0379, MMRM; Ratio = 0.77, 95% CI 2-sided [0.60 to 0.98], Standard Error of Mean 0.094

14. Post Hoc Outcome: Mean Group Difference in 10 Meter Walk/ Run
Description: Post-hoc analyses comparing the mean clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group.
  The 10-meter walk/run test is a performance measure used to assess walking speed in seconds over a short distance. It can be used as an assessment of functional mobility.
Time Frame: 20 weeks
Measure: Mean (Full Range); unit: Seconds
Groups:
- Cmax Lower Quantiles: Patients who showed lower exposure levels to tideglusib
- Cmax Upper Quantiles: Patients who showed higher exposure levels to tideglusib (50th percentile)
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 10 | 12 | 23
Seconds | 9.1 [6.9 to 16.1] | 8.7 [6.5 to 12.2] | 8.5 [3.9 to 18.7]

15. Post Hoc Outcome: Mean Change From Baseline Group Difference in 10 Meter Walk/ Run
Description: Post-hoc analyses comparing the mean change from baseline from clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group.
  The 10-meter walk/run test is a performance measure used to assess walking speed in seconds over a short distance. It can be used as an assessment of functional mobility.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 10 | 12 | 23
Seconds | 0.4 (1.7) | -1.5 (2.2) | -0.1 (1.8)
Statistical Analysis 1: Comparison: Cmax Upper Quantiles; Cmax upper quantiles group compared to the placebo group for mean change from baseline; two-tailed t-test assuming unequal variance; Test type: Superiority; p = 0.078, t-test, 2 sided

16. Post Hoc Outcome: Mean Group Difference in Peabody Picture Vocabulary Test (PPVT)
Description: Post-hoc analyses comparing the mean clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group. The PPVT-4 scale is a norm-referenced instrument for measuring the receptive (hearing) vocabulary. It contains training items and 228 test items, each consisting of four full-color pictures as response options on a page. Each test produces a raw score and a standard score. The raw score counts the number of correct responses. Raw scores are reported here as standardized scores are considered less appropriate for a pediatric population with cognitive deficits. Higher scores mean a better performance/receptive vocabulary. The lowest possible raw score is 0, the maximum raw score depends on the number of items administered so theoretically, the highest score possible on this test would be 228.
Time Frame: Baseline and week 20
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 9 | 9 | 19
score on a scale | 109 [35 to 185] | 134 [53 to 192] | 130 [51 to 191]

17. Post Hoc Outcome: Mean Change From Baseline Group Difference in Peabody Picture Vocabulary Test (PPVT)
Description: Post-hoc analyses comparing the mean change from baseline clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group. The PPVT-4 scale is a norm-referenced instrument for measuring the receptive (hearing) vocabulary. It contains training items and 228 test items, each consisting of four full-color pictures as response options on a page. Each test produces a raw score and a standard score. The raw score counts the number of correct responses. Raw scores are reported here as standardized scores are considered less appropriate for a pediatric population with cognitive deficits. Higher scores mean a better performance/receptive vocabulary. The lowest possible raw score is 0, the maximum raw score depends on the number of items administered so theoretically, the highest score possible on this test would be 228.
Time Frame: Baseline to week 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 9 | 9 | 19
score on a scale | 3 (14) | 6 (17) | -2 (10)
Statistical Analysis 1: Comparison: Cmax Upper Quantiles; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.29, t-test, 2 sided

18. Post Hoc Outcome: Mean Group Difference in Creatine Phosphokinase
Description: Post-hoc analyses comparing the mean clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group.
  Concentration of Creatine Phosphokinase (UI/L).
Time Frame: 20 weeks
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 11 | 12 | 23
IU/L | 147 [77 to 273] | 195 [42 to 460] | 299 [57 to 987]

19. Post Hoc Outcome: Mean Change From Baseline Group Difference in Creatine Phosphokinase
Description: Post-hoc analyses comparing the mean change from baseline in clinical responses of subjects with tideglusib exposures above the 50th percentile (who achieved the desired target exposure) with those subjects who showed lower exposure levels, and with the placebo group.
  Concentration of Creatine Phosphokinase (UI/L).
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: UI/L
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 11 | 12 | 23
UI/L | -17 (27) | -65 (147) | 30 (138)
Statistical Analysis 1: Comparison: Cmax Upper Quantiles; Cmax upper quantiles group compared to the placebo group for mean change from baseline (absolute value); two-tailed t-test assuming unequal variance; Test type: Superiority; p = 0.077, t-test, 2 sided

20. Post Hoc Outcome: Mean Group Difference in MDRI
Description: Post-hoc analyses comparing the mean clinical responses of subjects above and below the 50th percentile of tideglusib exposure levels with the placebo group. A multi-domain responder index (MDRI) analysis was performed by combining 5 objective endpoints. For each of the 5 endpoints, subjects were scored +1 point if their change exceeded or was equal to the threshold in a beneficial direction, -1 point if their change exceeded or was equal to the threshold in a detrimental direction and 0 points otherwise. The sum of these 5 scores were added together to provide an MDRI score between -5 and 5, where a higher score indicates greater overall improvement.
Time Frame: Baseline and week 20
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cmax Lower Quantiles | Cmax Upper Quantiles | Placebo
Number analyzed (Participants) | 11 | 12 | 23
score on a scale | 0.8 [-1.0 to 3.0] | 0.9 [-2.0 to 4.0] | -0.2 [-2.0 to 3.0]
Statistical Analysis 1: Comparison: Cmax Upper Quantiles; Cmax upper quantiles group compared to placebo group for mean Raw Score; two-tailed t-test assuming unequal variance; Test type: Superiority; p = 0.071, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Consent to end of study, up to 28 weeks
Description: A participant assigned to placebo was found to have some tideglusib levels (due to inadvertent exposure between siblings in opposing arms), and was therefore, included in the safety analysis and full analysis sets for tideglusib.
Arm/Group | Tideglusib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/25
Other Adverse Events (participants affected / at risk) | 20/28 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tideglusib (N=28) | Placebo (N=25)
Scoliosis Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tideglusib (N=28) | Placebo (N=25)
Nasopharyngytitis (Infections and infestations) | 3 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 2 (3) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to publish study results from his/her specific site. However, any publication that includes AMO Pharma confidential information cannot be submitted for publication without AMO Pharma's prior written approval.

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT03692312/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03692312/SAP_001.pdf